CLINICAL TRIAL: NCT04412694
Title: The Impact of Preoperative Oral Dexamethasone Supplementation on the Biochemical Parameters and Results of Surgical Treatment in Patients With Nontoxic Multinodular Goiter Undergoing Total Thyroidectomy.
Brief Title: The Effect of Preoperative Oral Dexamethasone Supplementation on the Outcome of Thyroidectomised Patients.
Acronym: Dexa
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Lodz (Other)
Responsible Party: Principal Investigator, Anna Grzegory, Principal Investigator, Medical University of Lodz
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MULODZ nr RNN/133/20/KE
Record Dates: First submitted 2020-05-23; First posted 2020-06-02 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2022-02

CONDITIONS: Hypocalcemia; Vitamin D Deficiency; Postoperative Complications; Postoperative Nausea; Postoperative Pain; Voice Hoarseness; Hypoparathyroidism Postprocedural
Keywords: dexamethasone; hypocalcaemia; hypocalcemic symptoms; postoperative complications; vitamin D deficiency; cytokines; postoperative pain; postoperative nausea; postoperative vomiting; hoarseness; acute phase proteins; hypoparathyroidism
MeSH Terms: conditions — Hypocalcemia; Vitamin D Deficiency; Postoperative Complications; Postoperative Nausea and Vomiting; Pain, Postoperative; Hoarseness; Hypoparathyroidism | interventions — Dexamethasone; Dietary Supplements; Sweetening Agents; Hematologic Tests; Thyroidectomy

STUDY DESIGN:
Intervention Model Description: Patients will be randomly assigned (coin toss) to the supplementation group (preoperative oral supplementation of dexamethasone (8mg in one dose) taken one hour before surgery) and to the placebo group (preoperative oral supplementation of sweetener taken one hour before surgery).
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- supplementation group (Experimental): Patients will receive preoperative oral supplementation of 8mg of dexamethasone (Dexamethasone Krka tablets (8mg), Warsaw, Poland) in a single dose taken once one hour before surgery. At 6 and 24 hour after surgery, clinical and laboratory parameters will be measured and evaluated.
  Interventions: Drug: Dexamethasone oral tablet 8mg (Dexamethasone Krka tablets(8mg), Warsaw, Poland).; Diagnostic Test: Preoparative blood laboratory tests; Diagnostic Test: Postoperative laboratory blood tests at 6 hour; Diagnostic Test: Postoperative laboratory blood tests at 24 hour; Diagnostic Test: Postoperative laboratory drainage fluid tests at 24 hour; Procedure: Total thyroidectomy; Other: Symptomatic hypocalcaemia at 6 hour; Other: Symptomatic hypocalcaemia at 24 hour; Other: Postoperative pain at 6 hour; Other: Postoperative pain at 24 hour; Other: Postoperative nausea and vomiting at 6 hour; Other: Postoperative nausea and vomiting at 24 hour; Other: Postoperative sore throat and hoarseness at 6 hour
- placebo group (Placebo Comparator): Patients will receive preoperative oral supplementation of sweetener (Clio tablets, sweetener with a dispenser, Instantina GES, Vienna, Austria) taken once in a single dose one hour before surgery. At 6 and 24 hour after surgery, clinical and laboratory parameters will be measured and evaluated.
  Interventions: Drug: Placebo oral sweetener (Clio tablets, sweetener with a dispenser, Instantina GES, Vienna, Austria).; Diagnostic Test: Preoparative blood laboratory tests; Diagnostic Test: Postoperative laboratory blood tests at 6 hour; Diagnostic Test: Postoperative laboratory blood tests at 24 hour; Diagnostic Test: Postoperative laboratory drainage fluid tests at 24 hour; Procedure: Total thyroidectomy; Other: Symptomatic hypocalcaemia at 6 hour; Other: Symptomatic hypocalcaemia at 24 hour; Other: Postoperative pain at 6 hour; Other: Postoperative pain at 24 hour; Other: Postoperative nausea and vomiting at 6 hour; Other: Postoperative nausea and vomiting at 24 hour; Other: Postoperative sore throat and hoarseness at 6 hour; Other: Postoperative sore throat and hoarseness at 24 hour

INTERVENTIONS:
Drug: Dexamethasone oral tablet 8mg (Dexamethasone Krka tablets(8mg), Warsaw, Poland). — Preoperative oral dexamathasone supplementation in a single dose of 8mg.
  Other Names: Supplementation
  Arms: supplementation group
Drug: Placebo oral sweetener (Clio tablets, sweetener with a dispenser, Instantina GES, Vienna, Austria). — Preoperative oral supplementation of sweetener in a single dose.
  Other Names: Placebo
  Arms: placebo group
Diagnostic Test: Preoparative blood laboratory tests — Preoperative parameters such as blood count, calcium, inorganic phosphates, albumin, alkaline phosphatase, C reactive protein, procalcitonin, 25-hydroxyvitamin D, fibrinogen, parathormone, magnesium, interleukin 1β, interleukin 6, interleukin 10, thyroid stimulating hormone, free thyroxine, free triiodothyronin will be measured in serum.
  Other Names: preoperative blood test
Diagnostic Test: Postoperative laboratory blood tests at 6 hour — At 6 hour after surgery such parameters as blood count, calcium, inorganic phosphates, albumin, alkaline phosphatase, C reactive protein, procalcitonin, 25-hydroxyvitamin D, fibrinogen, parathormone, magnesium will be measured in serum.
  Other Names: blood tests 6 hour
Diagnostic Test: Postoperative laboratory blood tests at 24 hour — At 24 hour after surgery such parameters as blood count, calcium, inorganic phosphates, albumin, alkaline phosphatase, C reactive protein, procalcitonin, 25-hydroxyvitamin D, fibrinogen, parathormone, magnesium, interleukin 1β, interleukin 6, interleukin 10 will be measured in serum.
  Other Names: blood tests 24 hour
Diagnostic Test: Postoperative laboratory drainage fluid tests at 24 hour — At 24 hour after surgery such parameters as interleukin 1β, interleukin 6, interleukin 10 will be measured in drainage fluid.
  Other Names: drainage fluid tests 24 hour
Procedure: Total thyroidectomy — Patients will undergo total thyroidectomy under general anesthesia.
  Other Names: thyroidectomy
Other: Symptomatic hypocalcaemia at 6 hour — At 6 hour after surgery patients will be assessed for signs of hypocalcaemia.
  Other Names: symptoms 6 hour
Other: Symptomatic hypocalcaemia at 24 hour — At 24 hour after surgery patients will be assessed for signs of hypocalcaemia.
  Other Names: symptoms 24 hour
Other: Postoperative pain at 6 hour — At 6 hour after surgery the incidence and intensity of postoperative pain will be evaluated according to Visual Analogue Scale (VAS).
  Other Names: pain 6 hour
Other: Postoperative pain at 24 hour — At 24 hour after surgery the incidence and intensity of postoperative pain will be evaluated according to Visual Analogue Scale (VAS).
  Other Names: pain 24 hour
Other: Postoperative nausea and vomiting at 6 hour — At 6 hour after surgery the incidence and intensity of postoperative nausea and vomiting will be evaluated.
  Other Names: nausea 6 hour
Other: Postoperative nausea and vomiting at 24 hour — At 24 hour after surgery the incidence and intensity of postoperative nausea and vomiting will be evaluated.
  Other Names: nausea 24 hour
Other: Postoperative sore throat and hoarseness at 6 hour — At 6 hour after surgery the incidence and intensity of postoperative sore throat and hoarseness will be evaluated.
  Other Names: hoarseness 6 hour
Other: Postoperative sore throat and hoarseness at 24 hour — At 24 hour after surgery the incidence and intensity of postoperative sore throat and hoarseness will be evaluated.
  Other Names: hoarseness 24 hour
  Arms: placebo group

SUMMARY:
Glucocorticoids are well known for their analgesic, anti-inflammatory, immunomodulatory and anti-emetic effects. Recovery time after thyroid surgery may depend on several factors, such as postoperative pain, nausea and vomiting, postoperative sore throat, voice disorders and symptomatic hypocalcaemia (low serum calcium level). However, there is little information in the literature about the preventive use of glucocorticosteroids in patients undergoing thyroid surgery. The aim of the study is to evaluate the clinical impact of preoperative oral dexamethasone supplementation on the surgical outcome in patients with multinodular goiter undergoing total thyroidectomy. Patients will be assigned to the supplementation group and the placebo group. In the supplementation group 8mg of dexamethasone will be administered orally one hour before surgery. In the postoperative period, the frequency and intensity of pain, nausea, vomiting, sore throat and hoarseness will be assessed. The incidence of symptoms of hypocalcaemia will also be evaluted. Preoperative and postoperative levels of vitamin D, cytokines, acute phase proteins and substances related to calcium metabolism will be measured in the blood. Cytokines levels in drainage fluid will also be assessed. The main hypothesis of the study is that in patients with supplementation postoperative discomfort and decrease in serum calcium and parathormone level and hypocalcemic symptoms will be less severe and the levels of proinflammatory substances will be decreased.

DETAILED DESCRIPTION:
Recovery time after thyroid surgery may depend on several factors, such as postoperative pain, nausea and vomiting, postoperative sore throat, phonation disorders associated with recurrent laryngeal nerve palsy, and symptomatic postoperative hypocalcaemia associated with postoperative hypoparathyroidism.

Glucocorticoids are well known for their analgesic, anti-inflammatory, immunomodulatory and anti-emetic effects. However, there is little information in the literature on the prophylactic use of glucocorticosteroids in patients undergoing thyroid surgery. In some previous studies, preoperative intravenous dexamethasone supplementation was associated with a reduced incidence of postoperative laryngeal nerve palsy, postoperative hypoparathyroidism, and with less severe postoperative pain, postoperative sore throat, nausea and vomiting. Patients receiving supplementation also had decreased levels of inflammatory biochemical parameters and proinflammatory cytokines.

Vitamin D deficiency is widespread in Poland. Vitamin D status has an impact on the postoperative complications in surgical patients. In previous study serum 25-hydroxyvitamin D is also suggested as a negative acute phase reactant, which has implications for acute and chronic inflammatory diseases. According to the authors, serum 25-hydroxyvitamin D level is an unreliable biomarker of vitamin D status after acute inflammatory insult.

In the early stages of inflammation, phagocytic cells and endothelium secrete proinflammatory cytokines, which include: interleukins: IL-1 α / β, IL-6, IL-8, TNF. The antagonistic group is anti-inflammatory cytokines, which include interleukins: IL-4, -5, -10, -13, produced by Th2 lymphocytes. These cytokines reduce the amount of interleukins secreted by Th1 lymphocytes.

Changes in the levels of proinflammatory and anti-inflammatory cytokines in the postoperative period were found in studies related to the assessment of surgical trauma. Pro-inflammatory interleukin 1 and interleukin 6 play an important role in many biological processes such as inflammation, sepsis and wound healing. Interleukin 6 expression is proportional to the extent of the surgical trauma. In turn, interleukin 10 is known as a cytokine that inhibits cytokine synthesis. Is one of the strongest immunosuppressive agents.

The aim of my study is to evaluate the impact of preoperative oral dexamethasone supplementation on the biochemical parameters and results of surgical treatment in patients with nontoxic multinodular goiter undergoing total thyroidectomy.

Patients admitted to the Department of General and Oncological Surgery, Medical University of Lodz with preoperative diagnosis of nontoxic multinodular goitre undergoing total thyroidectomy will be inculded to the study.

After obtaining written informed consent from all participants during a preoperative visit, they will be randomized to the supplementation group and the placebo group. The study will be a prospective, placebo-controlled and double-blind (for patient and surgeon) research.

Intervention: In the supplementation group a single dose of 8mg of dexamethasone will be given orally one hour before surgery (Dexamethasone Krka tablets (8mg), Warsaw, Poland). In the placebo group patients will receive a single tablet of sweetener one hour before operation (Clio tablets, sweetener with a dispenser, Instantina GES, Vienna, Austria).

Preoperatively in the group of all enrolled patients (in the supplementation group and in the placebo group) following tests will be measured in serum: blood count, calcium, inorganic phosphates, albumin, alkaline phosphatase, C reactive protein, procalcitonin, 25-hydroxyvitamin D, fibrinogen, parathormone, magnesium, interleukin 1β, interleukin 6, interleukin 10, thyroid stimulating hormone, free thyroxine, free triiodothyronine.

Total thyroidectomies with routine identification of the recurrent laryngeal nerves and parathyroid glands via a transverse cervicotomy under general anaesthesia will be performed by 3 experienced surgeons.

During the total thyroidectomy the number of parathyroid glands found intraoperatively will be registered.

At 6 hour after surgery in the group of all enrolled patients following tests will be measured in serum: blood count, calcium, inorganic phosphates, albumin, alkaline phosphatase, C reactive protein, procalcitonin, 25-hydroxyvitamin D, fibrinogen, parathormone, magnesium. In addiction, at 6 hour after surgery the incidence and intensity of symptomatic hypocalcaemia, postoperative pain (according to VAS scale), postoperative nausea and vomiting, postoperative sore throat and hoarseness will be evaluated.

At 24 hour after surgery in the group of all enrolled patients following tests will be measured in serum: blood count, calcium, inorganic phosphates, albumin, alkaline phosphatase, C reactive protein, procalcitonin, 25-hydroxyvitamin D, fibrinogen, parathormone, magnesium, interleukin 1β, interleukin 6, interleukin 10. Additionally, the level of interleukin 1β, interleukin 6 and interleukin 10 will be evaluated in drainage fluid. In addiction, at 24 hour after surgery the incidence and intensity of symptomatic hypocalcaemia, postoperative pain (according to Visual Analogue Scale - VAS scale), postoperative nausea and vomiting, postoperative sore throat and hoarseness will be evaluated.

The laboratory parameters will be determined by electrochemiluminescence on the Cobas E411 analyzer and spectrophotometric method on the AU680, Beckman Coulter analyzer. 25-hydroxyvitamin D levels will be measured using the chemiluminescent microparticle immunoassay (CMIA) (Architect 25-OHD). Interleukins levels will be determined by enzyme immunoassay method (EIA) (DGR Medtek) on ElizaMat 2 X analyzer.

Hypocalcemic symptoms will be categorized as mild (a tingling sensation and numbness of the hands or feet and perioral numbness) or severe (a positive Chvostek sign, Trousseau sign, tetany, and carpopedal spasms).

Postoperative hypocalcaemia will be defined as corrected calcium levels <2.0 mmol/l, even if recorded in one measurement only.

In both groups participants who will develop postoperative hypoparathyroidism (parathormone level <1.6 pmol/l at 6 or 24 hour after surgery) or symptomatic hypocalcaemia during hospitalisation will be treated with oral calcium (3 g/d - taken 1 g every 8 hours) and vitamin D derivatives (1 ug/d alfacalcidol taken once).

Intravenous calcium gluconate will be administered if symptoms persist despite oral supplementation.

Patients with symptomatic hypocalcaemia will receive supplementation until the symptoms subside. The treatment will be extended to 6 weeks in patients with hypoparathyroidism on the day of discharge.

The data will be statistically analysed. The main hypothesis of the study is that in patients with supplementation postoperative discomfort and decrease in serum calcium and parathormone level and hypocalcemic symptoms will be less severe and the levels of proinflammatory substances will be decreased. Vitamin D deficiency is probably common in operated patients and postoperative 25-hydroxyvitamin D levels are lower than those measured preoperatively.

The use of oral dexamethasone might be an effective strategy of prevention of complications after total thyroidectomy.

To the best of our knowledge, this is a pioneering study assessing the usefulness of preventive oral dexamethasone supplementation before total thyroidectomy in homogeneous group of patients with nontoxic multinodular goiter undergoing total thyroidectomy.

ELIGIBILITY:
Inclusion Criteria:

* patient's consent
* adult patients
* preoperative diagnosis of nontoxic multinodular goiter
* total thyroidectomy

Exclusion Criteria:

* lack of patient's consent
* hyperthyroidism currently or in the past
* retrosternal goiter
* thyroid malignanacy or suspected malignant thyroid tumor
* parathyroids disease
* malingant tumor in any location currently or in the past
* state after neck surgery
* state after radiotherapy
* bone diseases, osteoporosis
* sarcoidosis
* liver failure, hepatitis
* kidney stones, kidney failure (eGFR<60ml/min/1.73m2)
* taking nonsteroidal anti-inflammatory drugs
* steroid treatment
* stomach and duodenal ulcer disease currently or in the past
* active infection at the time of the study
* history of tuberculosis
* a period of 8 weeks before and 2 weeks after administration of the live vaccine
* unregulated hypertension
* diabetes
* psychiatric disorders
* glaucoma
* corneal ulcers or corneal injuries
* severe heart failure
* pheochromocytoma
* myasthenia gravis
* epilepsy
* head injury
* ulcerative colitis
* diverticulitis
* pregnancy
* breast-feeding
* hypokalaemia
* galactose intolerance
* lactase deficiency
* dexamethasone allergy, allergic to lactose, allergic to gelatinized starch, allergic to corn starch, allergic to colloidal anhydrous silica, allergic to magnesium stearate
* allergic reaction to substances contained in the sweetener: sodium cyclamate, sodium saccharin, sodium bicarbonate, sodium citrate.
* taking medications that affect calcium metabolism: anti-resorptive drugs, anabolic drugs, bisphosphonates, systemic glucocorticosteroids, thiazide diuretics, furosemide, proton pump inhibitors, antacids containing magnesium or aluminum salts, cholestyramine, colestipol, paraffin oil, salicylates, estrogen-containing oral contraceptives (hormonal contraceptives) , preparations containing calcium salts (regular intake), preparations of vitamin D or its analogues (regular intake)
* taking medications that increase the side effect of dexamethasone or enter into drug interactions with dexamethasone: acetazolamide, loop diuretics, thiazide diuretics, diuretics, amphotericin B, glucocorticosteroids, mineralocorticosteroids, tetracosactide and laxatives, carbenoxolone, chlorokine, hydroxychlorokine and meflocin, angiotensin converting enzyme inhibitors, thalidomide, cholinesterase inhibitors in patients with myasthenia gravis, fluorochonolones, ephedrine, barbiturates, rifabutin, rifampicin, phenytoin and carbamazepine, aminoglutethimide, bile acid binding resins, such as cholestyramine, antacids,activated carbon, antifungal azoles, ketoconazole, HIV protease inhibitors, macrolide antibiotics, estrogens, anti-tuberculosis drugs (isoniazid), cyclosporin, praziquantel, oral anticoagulants (coumarin), atropine and other anticholinergic drugs, somatotropin, protirel.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2022-09 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Postoperative hypocalcaemia | preoperatively and at 6 and 24 hour after surgery
  To evaluate the incidence of laboratory hypocalcaemia (corrected calcium serum level <2.0 mmol/l), the change in calcium levels and symptomatic hypocalcaemia in the postoperative period in the supplementation group and in the placebo group.
Postoperative hypoparathyroidism | preoperatively and at 6 and 24 hour after surgery
  To evaluate the incidence of hypoparathyroidism (parathormone serum level <1.6 pmol/l) and the change in parathormone levels in the postoperative period in the supplementation group and in the placebo group.

SECONDARY OUTCOMES:
Postoperative pain | at 6 and 24 hour after surgery
  To evaluate the intensity of postoperative pain according to Visual Analogue Scale (VAS scale) in the postoperative period in the supplementation group and in the placebo group. Minimum value is 0 (no pain) and maximum value is 10 (the worst possible pain). Higher scores mean a worse outcome.
Postoperative nausea on a verbal rating scale | at 6 and 24 hour after surgery
  To evaluate the incidence and the intensity of postoperative nausea in the postoperative period in the supplementation group and in the placebo group. The intensity of nausea will be rated on a verbal rating scale based on verbal responses of the patient to questions: 0 - no nausea; 1 - mild nausea (1 episode of nausea); 2 - moderate nausea (2 or 3 episodes of nausea ); and 3 - severe nausea (>3 episodes of nausea ). Higher scores mean a worse outcome.
Postoperative vomiting on a verbal rating scale | at 6 and 24 hour after surgery
  To evaluate the incidence and the intensity of postoperative vomiting in the postoperative period in the supplementation group and in the placebo group.The intensity of vomiting will be rated on a verbal rating scale based on verbal responses of the patient to questions: 0 - no episodes of vomiting; 1 - mild vomiting (1 episode of vomiting); 2 - moderate vomiting (2 or 3 episodes of vomiting); and 3 - severe vomiting (>3 episodes of vomiting).Higher scores mean a worse outcome.
Postoperative sore throat on a verbal rating scale | at 6 and 24 hour after surgery
  To evaluate the incidence and the intensity of postoperative sore throat in the postoperative period in the supplementation group and in the placebo group. Postoperative sore throat will be defined as discomfort at larynx or pharynx at rest and during swallowing after surgery. The intensity of sore throat will be rated on a verbal rating scale based on verbal responses of the patient to questions: 0 - none; 1 - mild sore throat (less severe than with a cold); 2 - moderate sore throat (similar with a cold); and 3 - severe sore throat (more severe than with a cold). Higher scores mean a worse outcome.
Postoperative hoarseness on a verbal rating scale | at 6 and 24 hour after surgery
  To evaluate the incidence and the intensity of postoperative hoarseness in the postoperative period in the supplementation group and in the placebo group. The intensity of hoarseness will be rated on a verbal rating scale based on verbal responses of the patient to questions: 0 - none; 1 - mild hoarseness (noticed by the patient only); 2 - severe hoarseness (obvious to observer); 3 - aphonia (silence of voice). Higher scores mean a worse outcome.

OTHER OUTCOMES:
Cytokines in serum | preoperatively and at 6 and 24 hour after surgery
  To evaluate the serum levels of cytokines such as interleukin 1β, interleukin 6, interleukin 10 and the change in cytokines levels in the postoperative period in the supplementation group and in the placebo group.
Cytokines in drain fluid | at 24 hour after surgery
  To evaluate the levels of cytokines such as interleukin 1β, interleukin 6, interleukin 10 in the drain fluid in the postoperative period in the supplementation group and in the placebo group.
Calcium phosphate homeostasis | preoperatively and at 6 and 24 hour after surgery
  To evaluate the serum levels of alkaline phosphatase,inorganic phosphates and magnesium and the change in their levels in the postoperative period in the supplementation group and in the placebo group.
Vitamin D | preoperatively and at 6 and 24 hour after surgery
  To evaluate the levels of 25-hydroxyvitamin D in the preoperative and postoperative period and the change in its levels in the supplementation group and in the placebo group. To evaluate the incidence of vitamin D deficiency in the group of operated patients.
Acute phase proteins | preoperatively and at 6 and 24 hour after surgery
  To evaluate the serum levels of albumin, C reactive protein, procalcitonin and fibrinogen and the change in their levels in the postoperative period in the supplementation group and in the placebo group.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Grzegory, MD, Principal Investigator — Medical University of Lodz, Poland
Locations (1):
- Department of General and Oncological Surgery, Medical University of Lodz, Lodz, Łódź Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Yes
All IPD will be included in planned publication.
Supporting Information: Study Protocol, SAP
Time Frame: starting 6 months after publication
Access Criteria: planned publication, journal website

REFERENCES:
- [Background] Schietroma M, Cecilia EM, Carlei F, Sista F, De Santis G, Lancione L, Amicucci G. Dexamethasone for the prevention of recurrent laryngeal nerve palsy and other complications after thyroid surgery: a randomized double-blind placebo-controlled trial. JAMA Otolaryngol Head Neck Surg. 2013 May;139(5):471-8. doi: 10.1001/jamaoto.2013.2821. PMID 23681030 (Retraction: PMID 30325981 JAMA Otolaryngol Head Neck Surg. 2018 Dec 1;144(12):1089)
- [Background] Yang C, Jung SM, Bae YK, Park SJ. The effect of ketorolac and dexamethasone on the incidence of sore throat in women after thyroidectomy: a prospective double-blinded randomized trial. Korean J Anesthesiol. 2017 Feb;70(1):64-71. doi: 10.4097/kjae.2017.70.1.64. Epub 2016 Nov 25. PMID 28184269
- [Background] Calkosinski I, Dobrzynski M, Calkosinska M, Seweryn E, Bronowicka-Szydelko A, Dzierzba K, Ceremuga I, Gamian A. [Characterization of an inflammatory response]. Postepy Hig Med Dosw (Online). 2009 Sep 3;63:395-408. Polish. PMID 19745226
- [Background] Waldron JL, Ashby HL, Cornes MP, Bechervaise J, Razavi C, Thomas OL, Chugh S, Deshpande S, Ford C, Gama R. Vitamin D: a negative acute phase reactant. J Clin Pathol. 2013 Jul;66(7):620-2. doi: 10.1136/jclinpath-2012-201301. Epub 2013 Mar 1. PMID 23454726
- [Background] Bennett NT, Schultz GS. Growth factors and wound healing: biochemical properties of growth factors and their receptors. Am J Surg. 1993 Jun;165(6):728-37. doi: 10.1016/s0002-9610(05)80797-4. PMID 8506974
- [Background] Gailit J, Clark RA. Wound repair in the context of extracellular matrix. Curr Opin Cell Biol. 1994 Oct;6(5):717-25. doi: 10.1016/0955-0674(94)90099-x. PMID 7530463
- [Background] Sakamoto K, Arakawa H, Mita S, Ishiko T, Ikei S, Egami H, Hisano S, Ogawa M. Elevation of circulating interleukin 6 after surgery: factors influencing the serum level. Cytokine. 1994 Mar;6(2):181-6. doi: 10.1016/1043-4666(94)90040-x. PMID 8032001
- [Background] Kalayci D, Dikmen B, Kacmaz M, Taspinar V, Ornek D, Turan O. [Plasma levels of interleukin-10 and nitric oxide in response to two different desflurane anesthesia flow rates]. Braz J Anesthesiol. 2014 Jul-Aug;64(4):292-8. doi: 10.1016/j.bjan.2013.06.009. Epub 2014 Jun 3. Portuguese. PMID 25096778
- [Background] Delogu G, Antonucci A, Signore M, Marandola M, Tellan G, Ippoliti F. Plasma levels of IL-10 and nitric oxide under two different anaesthesia regimens. Eur J Anaesthesiol. 2005 Jun;22(6):462-6. doi: 10.1017/s0265021505000797. PMID 15991511
- [Background] Turan A, Hesler BD, You J, Saager L, Grady M, Komatsu R, Kurz A, Sessler DI. The association of serum vitamin D concentration with serious complications after noncardiac surgery. Anesth Analg. 2014 Sep;119(3):603-612. doi: 10.1213/ANE.0000000000000096. PMID 25121616
- [Background] Pludowski P, Ducki C, Konstantynowicz J, Jaworski M. Vitamin D status in Poland. Pol Arch Med Wewn. 2016 Aug 9;126(7-8):530-9. doi: 10.20452/pamw.3479. Epub 2016 Aug 9. PMID 27509842